CLINICAL TRIAL: NCT00163839
Title: The Efficacy of a Pseudoallergen-Free Diet in the Treatment of Chronic Idiopathic Urticaria or Angioedema: A Randomised Controlled Study
Brief Title: The Efficacy of a Pseudoallergen-Free Diet in the Treatment of Chronic Idiopathic Urticaria and/or Angioedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 30/05; Ph: 00613 9276 3063
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2005-09

CONDITIONS: Urticaria; Angioedema
Keywords: Dietary Intervention; Pseudoallergen free diet
MeSH Terms: conditions — Urticaria; Angioedema | interventions — Diet Therapy

INTERVENTIONS:
Behavioral: Dietary Therapy

SUMMARY:
This study involves investigating the effects of a pseudoallergen-free (active) diet compared with a control (placebo) diet in the treatment of Chronic Idiopathic Urticaria (CIU) and/or Angioedema. The hypothesis is that over a four-week intervention period, the pseudoallergen-free diet will be more effective than the placebo diet in reducing the frequency and severity of CIU and/or Angioedema.

DETAILED DESCRIPTION:
The role of dietary pseudoallergens as a trigger for CIU and/or Angioedema is a controversial subject. 'Dietary Pseudoallergy' refers to the mimicking of IgE symptoms (such as rash, itch and swelling) by components of food in the absence of a true IgE mediated response (as diagnosed by RAST and skin prick testing).

The pseudoallergen-free diet excludes a range of naturally occuring chemicals (including salicylates, amines and brewers yeast) in addition to a range of artificial preservatives and additives (for example sulphites and glutamates). The control diet is based on the general dietary guidelines for the management of diabetes (including the principles of healthy eating, low glycemic index choices and a reduced saturated fat intake).

Subjects recruited into the study will have a 3 month history of CIU and/or Angioedema and will be randomly assigned to either the active or control arm of the study in a single blinded fashion. All subjects will be advised to cease antihistamine medication and will receive one-on-one dietary counselling by a Dietitian. The diet to which each subject has been assigned (ie either active or placebo) is to be followed for a 4 week duration. The frequency and severity of CIU and/or Angioedema as well as adherence to the diet are to be measured on both a daily and weekly basis by the subject via the completion of a clinical score card. The results of the score cards will be collated to determine the relative effects of each diet on these conditions.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Aged between 21 to 75 years
* 3 month history of Chronic Idiopathic Urticaria and/or Angioedema

Exclusion Criteria:

* age <21 and >75 years
* non english speaking
* systemic lupus erythematosis
* dysproteinemias
* thyrotoxicosis
* vasculitis
* infection

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-09

PRIMARY OUTCOMES:
The frequency and severity of CIU and/or angioedema (as determined via a five point rating scale)

SECONDARY OUTCOMES:
The relative use of antihistamines (ie how many, how often)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Connell, Masters, Principal Investigator — Alfred Hospital, Melbourne, Australia
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia